CLINICAL TRIAL: NCT05649215
Title: Low Back Activity Confidence Scale: Cross-cultural Adaptation, Reliability, and Validity of the Turkish Version
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Assistant Professor, Gazi University
Other Study IDs: 83116987-704
Record Dates: First submitted 2022-11-28; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Turkish version; Translation; Reliability; Validity
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Patients with low back pain
  Interventions: Other: No intervention will be applied.

INTERVENTIONS:
Other: No intervention will be applied. — This is a questionnaire study.

SUMMARY:
This study is aimed to carry out the Turkish version validity and reliability of the Low Back Activity Confidence Scale.

DETAILED DESCRIPTION:
Because self-efficacy represents a situation-specific construct and not a general or personality construct, confidence in performing one type of activity can differ significantly from confidence in performing other actions, all of which can contribute to a common outcome. Optimally, self-efficacy measures are tailored to assess individuals' confidence in exhibiting key behaviors related to recovery or alleviation from their own health condition or condition. Therefore, self-efficacy scales involve measuring an individual's confidence in each unique behavior or set of behaviors. Self-efficacy also explained more discomfort than pain intensity in patients with chronic pain. In addition, with appropriate insight and assessment, self-efficacy can perhaps be developed more effectively or appropriately than other non-modifiable (e.g. demographics) or less easily modifiable factors, such as fear beliefs and catastrophic thinking. Although several instruments have been developed to assess self-efficacy in low back pain, they do not address relevant functional and self-regulatory behaviors in the post-intervention clinical population. Therefore, the Low Back Activity Confidence Scale (LoBACS) was created to assess various forms of self-efficacy potentially related to low back pain. LoBACS is general, non-work-specific, but self-efficacy for backward functional activities such as standing, carrying, and pushing, self-regulation or self-control to manage one's thoughts, emotions, and behaviors to perform or avoid activities that may contribute to back health. and self-efficacy to do regular exercise, a core activity in a range of therapeutic interventions for low back pain. There is no Turkish version and validity study of LoBACS. This study is aimed to evaluate the validity and reliability of the Turkish version of LoBACS. The study of validity and reliability is planned with 104 individuals with low back pain. The sociodemographic characteristics of the individuals will be questioned by the investigators and then the patients will be evaluated with LoBACS, International Physical Activity Questionnaire (IPAQ), Back Pain Functional Scale (BPFS), Waddell Disability Index (WDI), Modified Oswestry Disability Index (MODI), Roland-Morris Disability Questionnaire (RMDQ), Short Form-36 (SF-36), Fear Avoidance Beliefs Questionnaire (FABQ) and Visual Analogue Scale (VAS). The test-retest will be re-administered by face-to-face interview technique after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* have any diagnosis of low back pain;
* who have had low back pain for at least 3 months;
* at least 18 years;
* to be able to read and write in Turkish;
* to volunteer.

Exclusion Criteria:

* poor knowledge of Turkish language;
* cognitive impairment;
* the presence of psychiatric limitations;
* chronic degenerative inflammatory or neurologic disorders;
* infections;
* systemic disorders;
* pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with low back pain between the ages of 18-60
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Low Back Activity Confidence Scale (LoBACS) | Two assessments- 7 minutes
  It was developed as a scale consisting of 15 items and 3 subscales in 2011 and was organized based on theoretical, rational distinctions and content. The functional self-efficacy subscale includes 7 items related to self-confidence for challenging functional activities (i.e. carrying, lifting, pushing, sitting, standing, walking, and climbing stairs), which are frequently mentioned for individuals with low back pain. The self-regulatory self-efficacy subscale includes 3 items related to confidence in caring for, controlling and coping with a back problem. Exercise self-efficacy subscale includes 5 items related to maintaining regular exercise for back health in different disability situations. Each item is evaluated on an 11-point scale ranging from 0% (no confidence) to 100% (full confidence), marked in 10% increments. A high score indicates a high level of confidence.
Back Pain Functional Scale (BPFS) | Single assessment- 7 minutes
  It is a scale that evaluates how much activity and functions of individuals are affected by their current low back pain complaints. Functions and activities evaluated in the scale; work, school, indoor activities, general habits, bending forward, wearing shoes/socks, lifting something from the ground, sleeping, sitting, standing, walking, going up/down stairs and driving. Individuals who do not drive can answer the last question as traveling. Each expression is scored between 0 and 5. The maximum score is 60 points, while the minimum score is 0. A score of 60 indicates that there is no difficulty in performance. The Turkish validity and reliability of the scale has been proven.
Waddell Disability Index (WDI) | Single assessment- 5 minutes
  It is used to evaluate the basic physical activities of daily life restricted by low back pain. It consists of 9 two-ended (yes/no) items, the total score is calculated by adding up the yes answers. The highest score of WDI is 9, and higher scores indicate more severe disability
Modified Oswestry Disability Index (MODI) | Single assessment- 5 minutes
  It includes 10 questions about pain intensity, personal care, lifting weights, walking, sitting, standing, sleeping, social life, travel and change in pain over time, each question has 6 options. The individual is asked to choose the one that best describes his/her situation from the options between 0 and 5 points in each question. The highest score is 50 points. An increase in the score indicates an increase in functional limitation, while a decrease in the score indicates an increase in functional level. According to the sum of the points, the evaluation is made as follows; 0 points: no functional disability, 1-10 points: mild functional disability, 11-30 points: moderate functional disability, 31-50 points: severe functional disability. The Turkish version, validity and reliability study was performed.
Roland Morris Disability Questionnaire (RMDQ) | Single assessment- 10 minutes
  It consists of 24 questions answered as 'Yes' or 'No'. 1 point is awarded for each yes answer and 0 for each no answer. The total score is found by adding the given points. The total score is between 0-24 values. High scores indicate a lack of physical activity. The Turkish version, validity and reliability study was performed.
International Physical Activity Questionnaire (IPAQ) | Single assessment- 5 minutes
  It is used to determine the physical activity levels of individuals. The short form consisting of 7 items divides the activity into different intensity levels as vigorous, moderate and walking. The time spent sitting is considered as a separate question. Turkish version, validity and reliability study was conducted in 2010.
Short Form-36 (SF-36) | Single assessment- 12 minutes
  It is one of the most common generic measures used to measure quality of life. This scale examines 8 dimensions of health, such as physical function, role limitations (due to physical and emotional problems), social function, mental health, vitality (energy), pain and general perception of health, with 36 items. While the maximum value of Short Form-36 is 100, its minimum value is 0. Increased scores indicate a better quality of life. As the score decreases, the quality of life worsens. The Turkish version, validity and reliability study of the scale was performed.
Fear Avoidance Beliefs Questionnaire (FABQ) | Single assessment- 5 minutes
  It is a questionnaire consisting of two sub-scales, physical activity and work activity, and 16 questions. The main purpose is to show the effect of activity-induced fear and avoidance belief on low back pain and disability. It is based on the strong relationship between increased fear avoidance belief and chronic disability due to low back pain. While the maximum value of Fear Avoidance Beliefs Questionnaire is 66, its minimum value is 0. In the evaluation, it is accepted that fear-avoidance behavior decreases as the total score approaches 0, and increases in fear-avoidance behavior as it approaches the maximum score. The Turkish version, validity and reliability study was performed.
Visual Analog Scale (VAS) | Single assessment- 1 minute
  It consists of a 10-centimeter straight line starting from 0 on the left to the right. A value of 0 is defined as "no pain" and a value of 10 as "worst pain". Individuals are instructed to draw a vertical line on the horizontal line that indicates where on the line the pain they are feeling is, and the length of the line is measured. The Turkish validity and reliability study of the VAS was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Halime ARIKAN, PhD, Study Chair — Tokat Gaziosmanpasa University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR